CLINICAL TRIAL: NCT04416672
Title: VIP: Validation of the Italian Version of the Patient-Reported Outcomes - Common Terminology Criteria for Adverse Events (PRO-CTCAE): A Prospective Multicenter Observational Study on Different Cancer Types
Brief Title: Validation of the Italian Version of the PRO-CTCAE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: VIP
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Malignant Neoplasms
Keywords: PRO-CTCAE; EORTC QLQ-C30 or Disease-Specific Questionnaire; HADS; PGIC Scale; Performance Status; Quality of Life
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PRO-CTCAE items — Enrolled patients will be asked to complete a subset of the PRO-CTCAE items based on cancer type, and the following instruments used as anchors to measure psychometric properties:
  * the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life disease-specific module, if a linguistically validated Italian version exists, or the General QLQ-C30, if the Italian version is not available.
  * the Hospital Anxiety and Depression Scale (HADS)
  * The Patients' Global Impression of Change (PGIC) Scale.

SUMMARY:
The aim of this study is to complete the validation process by testing the remaining two psychometric properties (validity and responsiveness) of the Italian version of the PRO-CTCAE in a large group of patients. In particular, for the first time this study will validate the tool for individual types of cancer and will provide information on psychometric properties based on the type of treatment used in clinical practice.

DETAILED DESCRIPTION:
This is a prospective observational study, conducted in Italian cancer centers located Nationwide.

The investigators plan to consider for validation 21tumor sites, which correspond to the conditions for which a specific EORTC module has been produced, plus all remaining cancer types classified as "other setting".

The study will take place during two planned visits, one the first the day of enrollment, the second after 3-6 weeks. Enrolled patients will be asked to complete a subset of the PRO-CTCAE items based on cancer type, and the following instruments used as anchors to measure psychometric properties:

* EORTC Quality of Life disease-specific module, if a linguistically validated Italian version exists, or the General QLQ-C30, if the Italian version is not available.
* the Hospital Anxiety and Depression Scale (HADS)
* The Patients' Global Impression of Change (PGIC) Scale

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of any type of cancer

  •≥18 years of age.
* Female or male
* With at least two planned clinic visits (a return visit within 3-6 weeks) to avoid the need of extra visits
* Actively receiving treatment for cancer (going to receive the second or further cycle)
* Any ECOG performance status (PS)
* Able to complete questionnaire by themselves or with assistance, by using a tablet
* Able to speak and understand Italian
* Providing informed written consent

Exclusion Criteria:

* Having any kind of psychiatric disorder or major cognitive dysfunction hampering the provision of informed consent.
* Having received more than 5lines of therapies
* Currently participating in other trials which imply the completion of Patient Reported Outcomes (PROs) in the same period
* Other important acute medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any type of cancer
Sampling Method: Probability Sample
Enrollment: 3675 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Validity of the italian version of the PRO-CTCAE | at baseline (up to 3weeks)
  Evaluation of the validity (degree to which an instrument accurately measures the underlying phenomenon) of single items of the PRO-CTCAE, Italian version, for each of the type of cancer considered
Validity of the italian version of the PRO-CTCAE | at 3 weeks (up to 6 weeks)
  Evaluation of the validity (degree to which an instrument accurately measures the underlying phenomenon) of single items of the PRO-CTCAE, Italian version, for each of the type of cancer considered
Responsiveness of the italian version of the PRO-CTCAE | at baseline (up to 3 weeks)
  Evaluation of responsiveness (ability of an instrument to show a change when there has been a change in the phenomenon) of single items of the PRO-CTCAE for each of the types of cancer considered.
Responsiveness of the italian version of the PRO-CTCAE | at 3 weeks (up to 6 weeks)
  Evaluation of responsiveness (ability of an instrument to show a change when there has been a change in the phenomenon) of single items of the PRO-CTCAE for each of the types of cancer considered.

SECONDARY OUTCOMES:
Differences in psychometric measures according to tumor type and treatment | at 3 weeks (up to 6 weeks)
  Evaluate any differences in psychometric measures according to:
  * type of cancer (breast, lung, liver ...)
  * type of treatment (chemotherapy, hormone therapy, immunotherapy, ...)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Perrone, MD, PhD, Principal Investigator — Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale
Locations (25):
- Italy (25):
  - Oncologia Medica per la Patologia Toracica- IRCCS Giovanni Paolo II, Bari
  - U.O.C. Oncologia Medica - Ospedale Senatore Antonio Perrino, Brindisi
  - Azienda Ospedaliero Universitaria di Cagliar, Cagliari
  - Oncologia Medica 2 - IRCCS AOU San Martino, Genova
  - Oncologia - A.O. Cardinale G. Panico, Lecce
  - Oncologia Medica - AO Vito Fazzi, Lecce
  - Oncologia Medica, Istituto Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - A.O.Ospedali Riuniti Papardo Piemonte U.O.C. di Oncologia Medica, Messina
  - Fondazione IRCCS, Istituto Nazionale dei Tumori, Milan
  - Ginecologia e Ostetricia - IRCCS Ospedale San Raffaele, Milan
  - Oncologia - ASST Rhodense - Presidio di Garbagnat, Milan
  - Oncologia - ASST Rhodense - Presidio di Rho, Milan
  - Istituto Nazionale Tumori, Dip. Uro-Ginecologico S.C. Oncologia Clinica Sperimentale Uro-Ginecologica, Naples
  - Oncologia Medica Toraco-Polmonare -Istituto Nazionale Tumori, Naples
  - Servizio di Oncologia Medica ed Ematologia - DAI di Internistica Polispecialistica- AOU Università degli studi della Campania "Luigi Vanvitelli", Naples
  - Struttura semplice Sarcomi ossa e tessuti molli, Istituto Nazionale Tumori, IRCCS, Fondazione G. Pascale, Naples
  - U.O.C. di Oncologia - Presidio Monaldi - AORN Ospedale dei Colli, Napoli
  - Istituto Oncologico Veneto, Padua
  - AOU Oncologia Medica, Parma
  - Oncologia traslazionale - ICS Maugeri di Pavia, Pavia
  - Oncologia Medica ed Ematologia, USL di Piacenza - Ospedale Guglielmo da Saliceto, Piacenza
  - Oncologia Medica 2 - Istituto Nazionale Tumori "Regina Elena", Roma
  - UOC Oncologia Medica 1 - Istituti Fisioterapici Ospitalieri - Istituto Nazionale Tumori Regina Elena, Roma
  - Oncologia - Ospedale S. G. Moscati, Taranto
  - Oncologia Medica - Istituto Sacro Cuore Don Calabria, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caminiti C, Maglietta G, Arenare L, Di Liello R, Migliaccio G, Barberio D, De Laurentiis M, Di Rella F, Nuzzo F, Pacilio C, Iodice G, Orditura M, Ciardiello F, Di Bella S, Cavanna L, Porta C, Giovanardi F, Ripamonti CI, Bilancia D, Aprile G, Ruelle T, Diodati F, Piccirillo MC, Iannelli E, Pinto C, Perrone F. Psychometric properties of patient-reported outcomes Common Terminology Criteria for adverse events (PRO-CTCAE(R)) in breast cancer patients: The prospective observational multicenter VIP study. Breast. 2024 Oct;77:103781. doi: 10.1016/j.breast.2024.103781. Epub 2024 Jul 20. PMID 39059033